CLINICAL TRIAL: NCT06804148
Title: MYVAL Transcatheter Heart Valve System - Prospective German Multicenter Registry
Acronym: German MYVAL S
Status: Recruiting | Type: Observational
Sponsor: Prof. Dr. med. Ingo Eitel (Other)
Responsible Party: Sponsor-Investigator, Prof. Dr. med. Ingo Eitel, Head of department of medical clinic II, University of Luebeck
Organization: University of Luebeck (Other)
Other Study IDs: 2024-500
Record Dates: First submitted 2025-01-27; First posted 2025-02-03 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Aortic Valve Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: Myval Transcatheter Heart Valve — The Myval TAVR bioprothesis is a balloon-expandable THV developed by Meril Lifesciences, which has novel operator friendly design features to improve deliverability and aid precise deployment.

SUMMARY:
Rational of the Myval THV - Prospective German Multicenter Registry is to evaluate the performance of this relatively new but very promising TAVR valve in a consecutive real-word, all-comers registry and to assess the long-term durability and efficacy of the Myval THV.

ELIGIBILITY:
Inclusion Criteria:

* Patient is going to be treated with Myval THV
* Age ≥ 18 years
* Ability to give informed consent

Exclusion Criteria:

* Pregnant and lactating women
* Patients with hyper sensitivity or allergy to aspirin, heparin, clopidogrel, ticlopidine, cobalt, nickel, chromium, molybdenum or any contrast media.
* Patients in whom anti-platelet and/or anticoagulant therapy are contra-indicated.
* Any condition, which in the Investigator's opinion, would preclude safe participation of patient in the registry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who will be treated with Myval TAVR are included in the registry.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2030-12-01 (Estimated); Study Completion 2030-12-30 (Estimated)

PRIMARY OUTCOMES:
It is a composite of: - All-cause mortality - All stroke - Moderate or severe paravalvular regurgitation | 5 Year

CONTACTS AND LOCATIONS:
Locations (1):
- Universitätsklinikum Schleswig-Holstein - Campus Lübeck, Lübeck, Schleswig-Holstein, Germany

IPD SHARING:
Plan to Share IPD: No